CLINICAL TRIAL: NCT03283735
Title: Deprescribing: a Portrait and Out-comes of the Reduction of Polypharmacy in Portugal
Acronym: DePil17-20
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Beira Interior (Other)
Responsible Party: Principal Investigator, Pedro Augusto Simões, Doctor, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UBIMED2017
Record Dates: First submitted 2017-09-08; First posted 2017-09-14 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Polypharmacy; Deprescriptions
Keywords: Deprescribing; Polypharmacy; Elderly; Enablement; Quality of Life

STUDY DESIGN:
Intervention Model Description: This phase of the study is expected to start in September 2019 and will last for 6 months.
  Two groups will be created with a minimum of 190 patients each, one of which will be composed from patients from the region of Aveiro, Coimbra and Guarda and the other from patients from the region of Castelo Branco, Leiria and Viseu. In the intervention group the investigators will give enablement tools and talks with their GPs about how to issue the problem of polypharmacy. The information given in this group will result from the knowledge obtained in phase II in the shape of small leaflets and other information materials to be made according to the best practice, to be given and remembered at scheduled times to the intervention group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderly Enablement (Experimental): The investigators will give enablement tools and talks with their GPs about how to issue the problem of polypharmacy.
  Interventions: Behavioral: Elderly Enablement
- Control (No Intervention): This will be the control group.

INTERVENTIONS:
Behavioral: Elderly Enablement — The information given in this group will result from the knowledge obtained in previous phase of the study in the shape of small leaflets and other information materials to be made according to the best practice, to be given and remembered at scheduled times to the intervention group
  Arms: Elderly Enablement

SUMMARY:
This study protocol comprises three phases. The first two phases will be nationwide and aim to evaluate the prevalence and patterns of polypharmacy and assess the barriers and facilitators of deprescribing perceived by older adults, as well as their willingness to be deprescribed and to self-medicate. The third and last phase will be a non-pharmacological randomised clinical study to measure the impact of enablement of older adults in their willingness to be deprescribed and related quality of life.

DETAILED DESCRIPTION:
Study design

This is a three-phase study:

1. Cross-sectional, analytical study of the prevalence and patterns of polypharmacy, namely sociodemographic and clinical profiles (age, genre, area of residence and years of study) and about medication (number of drugs and their active component), in older adults attending Primary Care in Portugal.
2. Cross-sectional, triangulation study of older adults' perception of Barriers to and Facilitators of Deprescribing, Willingness to be Deprescribed and Willingness to Self-medicate.
3. Non-pharmacological randomised clinical study of the impact of enablement of older adults in their willingness to be Deprescribed and related Quality of Life.

Phase I: prevalence of polypharmacy in older adults attending primary care in Portugal Design Cross-sectional, analytical study.

Setting: Primary Care Centres in Portugal will be randomly selected from the five main-land Portuguese Healthcare Administrative Regions and two Autonomous Regions (Madeira and Azores), in order to obtain a national geographical representative sample.

Sample size Since the prevalence of polypharmacy in older adults is unknown, the investigators used as base of population all older adults in Portugal. For the study, the investigators used a 95% confidence interval (CI) and a maximum precision error of 5%, so a minimum of 385 patients should be recruited.

Study procedures This phase of the study starts in November 2017. General Practitioners (GPs) sampling is made according to existing files of previous projects adherent GPs, in other epidemiological studies. After the selection of GPs, those who accept to participate will recruit their own patients. Assuming that a GP will be able to include at least 6 patients in a 3-week period, a total of 65 GPs will be enrolled in the study: 21 in North of Portugal (31.7%), 16 in Centre of Portugal (24.7%), 18 in Lisbon-Tejo Valley (27.4%), 5 in Alentejo (8.4%), 3 in Algarve (4.3%), 1 in Azores (1.6%) and 1 in Madeira (1.9%) in accordance with the distribution of Portuguese old adult population (≥65 years) in Portugal according with Pordata (www.pordata.pt).

Enrolled GPs will be instructed to collect all necessary data about their patients meeting the eligibility criteria.

Data collection The collection of the data will occur in November 2017. GPs will be responsible for collecting all data about patients' sociodemographic characteristics, as well as morbidity and medication, during their consultations.

Data will be electronically stored in a database specifically designed for this study using MS Access 2010. Data will be encrypted and password protected. Information will be treated in strict confidentiality to protect the privacy of patients. The investigators will have no access to the data of the patient, except the one provided by the GP meaning that the only person to know who is being studied is the GP.

Before the collection of data, there will be online reunions with the GPs participating in the study.

Statistical analysis A descriptive analysis will be performed to all study variables, namely the number of valid observations, mean±SD, median and range for quantitative variables and absolute and relative frequencies for qualitative variables. Prevalence of polypharmacy (considering definition: ≥5 drugs vs ≥ the median number) will be calculated together with corresponding 95% CI. Moreover, the prevalence of polypharmacy will be estimated by subgroups, namely age, gender, residence area and formal education. Univariate analysis will be conducted to study the associations between those characteristics and polypharmacy using χ2 test (qualitative characteristics) or t test/Mann-Whitney (quantitative characteristics). Multiple logistic regressions will be carried out considering the presence of polypharmacy as the dependent variable and patients' characteristics as the independent variables in order to calculate odds ratio (ORs) and corresponding 95% CI. Total number of drugs taken by patient and their pharmacological classes will also be summarised together with 95% CI, and multiple regressions may be performed to analyse its association with patients' characteristics. All tests will be two-sided using a significance level of 0.05. Statistical analysis will be conducted using SPSS V.23.0 or higher.

Phase II: patients' perception of barriers to and facilitators of deprescribing, willingness to be deprescribed and actual self-medication in adult patients with polypharmacy attending primary care in Portugal Objectives To assert reasons and facilitators, willingness to be deprescribed and actual self-medication

Design Cross-sectional, analytical study.

Setting It will be the same of the phase I.

Sample size A minimum of 385 patients will be included in phase II in order to obtain a sample with a 95% CI and a maximum precision error of 5%.

Study procedures This phase of the study is expected to start in June 2018. Again, GPs sampling will be made according to existing files and those who accept to participate will recruit their own patients. Patients from phase I can be enrolled in phase II. Assuming that a GP will be able to include at least 6 patients in a 3-week period, a total of 65 GPs has to be enrolled in the study, with the same distribution of the phase I. Enrolled GPs will be instructed to invite all patients meeting the eligibility criteria.

Data collection The collection of the data will occur in June 2018. Patient's socio-demographic and clinical characteristics and medication will be registered using the same methodology as described in phase I. The investigators will also collect outcome measures of some tests.

Statistical analysis Descriptive statistics will be computed for all variables together with 95% CI whenever relevant and applicable. Associations between qualitative-independent variables will be tested using χ2 test. Comparisons between two or more independent groups regarding a quantitative variable are to be conducted using analysis of variance (ANOVA) or Kruskal-Wallis non-parametric test, if normality assumption is not met. ANCOVA may also be used to adjust for potential confounding factors. Associations between quantitative independent variables will be analysed using Pearson's or Spearman's correlation coefficient depending on normality assumption. All tests will be two-sided, considering a significance level of 0.05.

Phase III: impact of enablement of older adults in their willingness to deprescribe and quality of life Design Non-pharmacological randomised clinical study, intended to last for six months.

Setting Primary Care Centres in Portugal will be randomly selected from six Health Centres of Centre of Portugal (Aveiro, Castelo Branco, Coimbra, Guarda, Leiria and Viseu)

Sample size Will be created two groups with a minimum of 190 patients each (one will be the intervention group and the other the control).

Study procedures This phase of the study is expected to start in September 2019 and will last for 6 months.

Again, GPs sampling will be made according to existing files and those who accept to participate will recruit their own patients. Patients from previous phases can be enrolled in phase III. Assuming that a GP will be able to include at least 6 patients, a total of 64 GPs has to be enrolled in the study. Enrolled GPs will be instructed to invite all patients meeting the eligibility criteria.

Two groups will be created with a minimum of 190 patients each, one of which will be composed from patients from the region of Aveiro, Coimbra and Guarda and the other from patients from the region of Castelo Branco, Leiria and Viseu. In the intervention group the investigators will give enablement tools and talks with their GPs about how to issue the problem of polypharmacy. The information given in this group will result from the knowledge obtained in phase II in the shape of small leaflets and other information materials to be made according to the best practice, to be given and remembered at scheduled times to the intervention group.

Data collection The collection of the data will occur in the beginning and end of phase II. Patient's socio-demographic and clinical characteristics and medication will be registered using the same methodology as described in phase I. The investigators will also collect outcome measures of applied tests.

Statistical analysis Descriptive statistics will be computed for all variables together with 95% CI whenever relevant and applicable. Associations between qualitative-independent variables will be tested using χ2 test. Comparisons between two or more independent groups regarding a quantitative variable are to be conducted using analysis of variance (ANOVA) or Kruskal-Wallis non-parametric test, if normality assumption is not met. ANCOVA may also be used to adjust for potential confounding factors. Associations between quantitative independent variables will be analysed using Pearson's or Spearman's correlation coefficient depending on normality assumption. All tests will be two-sided, considering a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending to the primary care consultation in the selected health centres.

Exclusion Criteria:

* Being acutely unwell in the last three weeks
* Refuse to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Willingness to be deprescribed after the intervention with open-questions | six months
  Assess the enablement of older adults while being Deprescribed in the rise of Willingness to be Deprescribed with two open-questions (one to assess the facilitators and the other to assess the barriers) together with their perception of medication (Beliefs about Medicines Questionnaire).

SECONDARY OUTCOMES:
Quality of life after the intervention with EQ-5D | six months
  Assess the enablement of older adults while being Deprescribed in the rise of their Quality wtih EuroQol Five Dimensions Questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Augusto Simões, Master, Principal Investigator — University of Beira Interior

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Machado-Alba JE, Gaviria-Mendoza A, Machado-Duque ME, Chica L. Deprescribing: a new goal focused on the patient. Expert Opin Drug Saf. 2017 Feb;16(2):111-112. doi: 10.1080/14740338.2017.1273347. Epub 2016 Dec 26. PMID 27984921
- [Background] Scott IA, Hilmer SN, Reeve E, Potter K, Le Couteur D, Rigby D, Gnjidic D, Del Mar CB, Roughead EE, Page A, Jansen J, Martin JH. Reducing inappropriate polypharmacy: the process of deprescribing. JAMA Intern Med. 2015 May;175(5):827-34. doi: 10.1001/jamainternmed.2015.0324. PMID 25798731
- [Background] Galazzi A, Lusignani M, Chiarelli MT, Mannucci PM, Franchi C, Tettamanti M, Reeve E, Nobili A. Attitudes towards polypharmacy and medication withdrawal among older inpatients in Italy. Int J Clin Pharm. 2016 Apr;38(2):454-61. doi: 10.1007/s11096-016-0279-4. Epub 2016 Mar 7. PMID 26951120
- [Background] Halvorsen KH, Selbaek G, Ruths S. Trends in potentially inappropriate medication prescribing to nursing home patients: comparison of three cross-sectional studies. Pharmacoepidemiol Drug Saf. 2017 Feb;26(2):192-200. doi: 10.1002/pds.4142. Epub 2016 Dec 9. PMID 27935150
- [Background] Sirois C, Ouellet N, Reeve E. Community-dwelling older people's attitudes towards deprescribing in Canada. Res Social Adm Pharm. 2017 Jul-Aug;13(4):864-870. doi: 10.1016/j.sapharm.2016.08.006. Epub 2016 Aug 31. PMID 27663392
- [Background] Sivagnanam G. Deprescription: The prescription metabolism. J Pharmacol Pharmacother. 2016 Jul-Sep;7(3):133-7. doi: 10.4103/0976-500X.189680. PMID 27651709
- [Background] Sluggett JK, Ilomaki J, Seaman KL, Corlis M, Bell JS. Medication management policy, practice and research in Australian residential aged care: Current and future directions. Pharmacol Res. 2017 Feb;116:20-28. doi: 10.1016/j.phrs.2016.12.011. Epub 2016 Dec 10. PMID 27965033
- [Background] Farrell B, Tsang C, Raman-Wilms L, Irving H, Conklin J, Pottie K. What are priorities for deprescribing for elderly patients? Capturing the voice of practitioners: a modified delphi process. PLoS One. 2015 Apr 7;10(4):e0122246. doi: 10.1371/journal.pone.0122246. eCollection 2015. PMID 25849568
- [Background] Scott IA, Anderson K, Freeman CR, Stowasser DA. First do no harm: a real need to deprescribe in older patients. Med J Aust. 2014 Oct 6;201(7):390-2. doi: 10.5694/mja14.00146. PMID 25296059
- [Background] Turner JP, Edwards S, Stanners M, Shakib S, Bell JS. What factors are important for deprescribing in Australian long-term care facilities? Perspectives of residents and health professionals. BMJ Open. 2016 Mar 10;6(3):e009781. doi: 10.1136/bmjopen-2015-009781. PMID 26966056
- [Background] Reeve E, Andrews JM, Wiese MD, Hendrix I, Roberts MS, Shakib S. Feasibility of a patient-centered deprescribing process to reduce inappropriate use of proton pump inhibitors. Ann Pharmacother. 2015 Jan;49(1):29-38. doi: 10.1177/1060028014558290. Epub 2014 Nov 10. PMID 25385826
- [Background] Reeve E, Wiese MD, Hendrix I, Roberts MS, Shakib S. People's attitudes, beliefs, and experiences regarding polypharmacy and willingness to Deprescribe. J Am Geriatr Soc. 2013 Sep;61(9):1508-14. doi: 10.1111/jgs.12418. Epub 2013 Aug 26. PMID 24028356
- [Background] Palagyi A, Keay L, Harper J, Potter J, Lindley RI. Barricades and brickwalls--a qualitative study exploring perceptions of medication use and deprescribing in long-term care. BMC Geriatr. 2016 Jan 15;16:15. doi: 10.1186/s12877-016-0181-x. PMID 26767619
- [Background] Reeve E, Low LF, Shakib S, Hilmer SN. Development and Validation of the Revised Patients' Attitudes Towards Deprescribing (rPATD) Questionnaire: Versions for Older Adults and Caregivers. Drugs Aging. 2016 Dec;33(12):913-928. doi: 10.1007/s40266-016-0410-1. PMID 27785734
- [Background] Reeve E, To J, Hendrix I, Shakib S, Roberts MS, Wiese MD. Patient barriers to and enablers of deprescribing: a systematic review. Drugs Aging. 2013 Oct;30(10):793-807. doi: 10.1007/s40266-013-0106-8. PMID 23912674
- [Background] Jansen J, Naganathan V, Carter SM, McLachlan AJ, Nickel B, Irwig L, Bonner C, Doust J, Colvin J, Heaney A, Turner R, McCaffery K. Too much medicine in older people? Deprescribing through shared decision making. BMJ. 2016 Jun 3;353:i2893. doi: 10.1136/bmj.i2893. No abstract available. PMID 27260319
- [Background] Reeve E, Shakib S, Hendrix I, Roberts MS, Wiese MD. Review of deprescribing processes and development of an evidence-based, patient-centred deprescribing process. Br J Clin Pharmacol. 2014 Oct;78(4):738-47. doi: 10.1111/bcp.12386. PMID 24661192
- [Background] Whitman AM, DeGregory KA, Morris AL, Ramsdale EE. A Comprehensive Look at Polypharmacy and Medication Screening Tools for the Older Cancer Patient. Oncologist. 2016 Jun;21(6):723-30. doi: 10.1634/theoncologist.2015-0492. Epub 2016 May 5. PMID 27151653
- [Background] Page AT, Clifford RM, Potter K, Schwartz D, Etherton-Beer CD. The feasibility and effect of deprescribing in older adults on mortality and health: a systematic review and meta-analysis. Br J Clin Pharmacol. 2016 Sep;82(3):583-623. doi: 10.1111/bcp.12975. Epub 2016 Jun 13. PMID 27077231
- [Background] Beer C, Loh PK, Peng YG, Potter K, Millar A. A pilot randomized controlled trial of deprescribing. Ther Adv Drug Saf. 2011 Apr;2(2):37-43. doi: 10.1177/2042098611400332. PMID 25083200
- [Background] Reeve E, Shakib S, Hendrix I, Roberts MS, Wiese MD. The benefits and harms of deprescribing. Med J Aust. 2014 Oct 6;201(7):386-9. doi: 10.5694/mja13.00200. PMID 25296058
- [Background] Ryan R, Hill S. Making rational choices about how best to support consumers' use of medicines: a perspective review. Ther Adv Drug Saf. 2016 Aug;7(4):159-64. doi: 10.1177/2042098616651198. Epub 2016 May 20. PMID 27493719
- [Background] Tannenbaum C, Martin P, Tamblyn R, Benedetti A, Ahmed S. Reduction of inappropriate benzodiazepine prescriptions among older adults through direct patient education: the EMPOWER cluster randomized trial. JAMA Intern Med. 2014 Jun;174(6):890-8. doi: 10.1001/jamainternmed.2014.949. PMID 24733354
- [Background] Reeve E, Low LF, Hilmer SN. Beliefs and attitudes of older adults and carers about deprescribing of medications: a qualitative focus group study. Br J Gen Pract. 2016 Aug;66(649):e552-60. doi: 10.3399/bjgp16X685669. Epub 2016 Jun 6. PMID 27266865
- [Background] Gnjidic D, Le Couteur DG, Kouladjian L, Hilmer SN. Deprescribing trials: methods to reduce polypharmacy and the impact on prescribing and clinical outcomes. Clin Geriatr Med. 2012 May;28(2):237-53. doi: 10.1016/j.cger.2012.01.006. Epub 2012 Feb 21. PMID 22500541
- [Derived] Simoes PA, Santiago LM, Simoes JA. Deprescribing in primary care in Portugal (DePil17-20): a three-phase observational and experimental study protocol. BMJ Open. 2018 Jul 17;8(7):e019542. doi: 10.1136/bmjopen-2017-019542. PMID 30018092

DOCUMENTS (1):
  • Study Protocol (2017-09-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT03283735/Prot_001.pdf